CLINICAL TRIAL: NCT02614417
Title: Sleep-disordered Breathing in Eisenmenger Syndrome
Status: Completed | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Cristel Sørensen, MD, Rigshospitalet, Denmark
Other Study IDs: 2012-01
Record Dates: First submitted 2015-09-28; First posted 2015-11-25 (Estimated); Last update posted 2015-11-25 (Estimated); Status verified 2015-11

CONDITIONS: Eisenmenger Syndrome; Congenital Heart Disease; Sleep-disordered Breathing
MeSH Terms: conditions — Eisenmenger Complex; Heart Defects, Congenital; Sleep Apnea Syndromes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Polysomnography: Patients undergo an one-night in-hospital polysomnography to diagnose sleep-disordered breathing
  Interventions: Other: Polysomnography

INTERVENTIONS:
Other: Polysomnography — One night polysomnography performed using standard techniques and scored in accordance with American Academy of Sleep Medicine standards. Polysomnography monitors sleep by electroencephalography (F4-A1, C4-M1, O2-M1 F3-M2, C3-M2, O1-A2), electro-myography (submental and tibialis anterior muscles), electro-oculography, nasal flow, respiratory effort, pulse oximetry and transcutaneous carbon dioxide partial pressure.

SUMMARY:
Sleep-disordered breathing (SDB) is a wellknown comorbidity in cardiovascular disease. Knowledge about SDB in adult congenital heart disease is limited.

DETAILED DESCRIPTION:
Congenital heart defects (CHD) occur in approximately 1% of all live births. Around 5% of adults with CHD develop pulmonary arterial hypertension (PAH), with 25-50% of these patients exhibiting the most serious form, Eisenmenger syndrome. Eisenmenger syndrome is caused by a systemic-to-pulmonary shunt, which eventually leads to high pulmonary vascular resistance with right-to-left or bi-directional shunt. Right-to-left shunting reduces the systemic arterial oxygen capacity and consequently causes cyanosis, which may result in hypoxic tissue damage and multi-organ disease.

The natural history of Eisenmenger syndrome (ES) is generally poor compared to the general population with the latest reported actual survival rates of 94%, 74% and 52% at 40, 50 and 60 years of age, respectively. Until recently conventional symptomatic treatment with diuretics, digitalis, antiarrhythmic, anticoagulants, iron supplement, oxygen therapy, and ultimately heart-lung transplantation were the only options. Most patients die from progressive cardiovascular disease and heart failure, sudden heart death or haemoptysis.

However, the introduction of advanced therapy (AT) has improved symptoms and may also have changed to prognosis of these patients. Thus, newer studies have shown beneficial effect of treatment with advanced therapy including endothelin receptor antagonists, phosphodiesterase-5 inhibitors, and prostanoids. These pulmonary vasodilators are now recognized as targeted therapy in Eisenmenger syndrome.

Sleep-disordered breathing (SDB) with predominantly obstructive or central sleep apnoea (OSA/CSA) with Cheyne-Stokes respiration (CSR) is shown to be a common comorbidity in patients with heart failure (HF), as it is present in at least 50 % of these patients. In the general Danish population the estimated prevalence is 3-18% in men and 5-7% in women.

Studies in HF patients also suggest an increased rate of central sleep apnoea (CSA) versus obstructive sleep apnoea (OSA) compared to the general population. SDB may promote the progression of chronic heart failure (HF) and is independently associated with a decreased survival rate.

The standard treatment for patients with OSA is nocturnal continuous positive airway pressure (CPAP) usually delivered with a tight fitting nasal mask. The benefits of CPAP are well established in this group of patients, as opposed to CSA-patients. The largest randomized study demonstrated no effect of nocturnal CPAP in patients with HF and CSA on heart transplant-free survival, but improvements in apnoea frequency, blood oxygenation and left ventricle function. While CPAP and other assisted breathing devices may be used in SDB related to HF, this have no place in the treatment of patients with ES, as any rise in the intra-thoracic pressure and consequently increased PVR and right-to-left shunting will worsen the cyanosis.

The treatment of CSA in HF remains controversial; however aggressive optimization of the medical treatment in congestive heart failure seems to improve the condition.

In these patients, the effect of CPAP, nocturnal oxygen and drugs stimulating the central respiratory drive are less well documented or related to adverse events such as increased risk of arrhythmias.

Though the relationship between HF and SDB is well established, the prevalence and influence of SDB in Eisenmenger syndrome has not previously been examined.

There are many similarities between ES and HF, but several important differences are also present. In congestive heart failure the ventricular insufficiency is related to an increased left side filling pressure followed by pulmonary stasis or oedema, whereas ES patients often have a normal filling pressure and normal systemic vascular resistance, but high pulmonary vascular resistance (PVR) and cyanosis due to the right-left shunt.

The aims of this study are to examine a group of Eisenmenger Syndrome patients to establish the prevalence of SDB in this patient group, to examine the mechanism (CSA or OSA) behind SDB in Eisenmenger syndrome, and to relate the presence of SDB to a higher level of secondary erythrocytosis.

If a role of SDB in ES is demonstrated, further studies will be necessary to demonstrate whether SDB in Eisenmenger syndrome can be altered by advanced therapy.

Hypotheses

* The prevalence of SDB in Eisenmenger syndrome is higher than in the general population.
* SDB in Eisenmenger syndrome is caused by a central rather than obstructive mechanism.
* SDB in Eisenmenger syndrome is related to a more pronounced secondary erythrocytosis than explained by a daytime measurement of oxygen saturation.

ELIGIBILITY:
Inclusion Criteria:

* Eisenmenger Syndrome (definition: Pulmonary ≥ systemic vascular resistance with pulmonary-to-systemic shunt and cyanosis (periphery oxygen saturation < 92% at rest and/or < 87% during exercise).
* Stable for ≥ 3 months (no hospitalization, no change of medication, no deterioration).

Exclusion Criteria:

* Down's syndrome.
* Iron deficiency (definition: Ferritin < 12 µg/l and/or transferring saturation < 20%).
* Regular phlebotomy.
* Suspicion of risk of non-compliance.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Eisenmenger syndrome
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2013-06; Primary Completion 2015-08 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Apnoea-hypopnoea index | 1 night on Day 1
  Prevalence of sleep-disordered breathing during 1 night polysomnography measured by apnoea-hypopnoea index.

SECONDARY OUTCOMES:
Sleep stages | 1 night on Day 1
  Characterize the sleep architecture during 1 night polysomnography by evaluating the time spend in various sleep stages (N1, N2, N3, REM, measured by EEG)